CLINICAL TRIAL: NCT00780494
Title: A Phase II Study of Capecitabine, Carboplatin, and Bevacizumab for Metastatic or Unresectable Gastroesophageal Junction and Gastric Adenocarcinoma
Brief Title: Ph II of Capecitabine, Carboplatin & Bevacizumab for Gastroesophageal Junction & Gastric Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-11911; 98587 (Other: Stanford University Alternate IRB Approval Number); SU-07082008-1238 (Other: Stanford University); GI0002 (Other: OnCore); IRB-11911 (Other: Stanford IRB)
Record Dates: First submitted 2008-10-23; First posted 2008-10-27 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Stomach Cancer; Gastric (Stomach) Cancer; Neoplasm of Cardioesophageal Junction; Gastrointestinal Stromal Tumor (GIST)
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Stromal Tumors | interventions — Bevacizumab; Carboplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- bevacizumab+ carboplatin +capecitabine (Experimental): Participants receive bevacizumab 15 mg/kg intravenously followed by carboplatin AUC 6 intravenously on Day 1 of a 21-day cycle, concurrently with capecitabine 850 mg/m2 twice-daily by mouth on Cycle Days 1-to-14, followed by a 1-week break.
  Interventions: Drug: bevacizumab; Drug: carboplatin; Drug: capecitabine

INTERVENTIONS:
Drug: bevacizumab — Intravenous 15 mg/kg
  Other Names: Avastin
Drug: carboplatin — AUC 6, Intravenously Day 1 every 21 days
  Other Names: Paraplatin
Drug: capecitabine — 850mg/m2, Orally twice daily days 1-14 every 21 days.
  Other Names: Xeloda

SUMMARY:
To investigate bevacizumab in combination with carboplatin and capecitabine for patients with unresectable or metastatic GEJ or gastric cancers. We hope that by adding bevacizumab to standard chemotherapy for this patient population we will improve Progression Free Survival by 90% over historical controls.

DETAILED DESCRIPTION:
Primary Objectives:

To investigate if the addition of Bevacizumab to standard chemotherapy for metastatic or unresectable GEJ and gastric adenocarcinoma will improve PFS by 90% over historical controls.

Secondary Objectives:

* Assess toxicities using CTCAE v3.0
* Evaluate overall survival (OS) using Kaplan-Meier analysis
* Evaluate objective response rate (RR) by RECIST criteria
* Explore biomarkers of tumor response: CEA, CA 19.9, and serum VEGF
* Bank serum and tissue for future correlative studies
* Evaluate CT Perfusion to predict early therapeutic response to combination chemotherapy and anti-angiogenic therapy (OPTIONAL).

ELIGIBILITY:
Inclusion Criteria:

Subjects must be treated at Stanford University Medical Center for the entire length of study participation.

1. Patients with histologically or cytologically confirmed adenocarcinoma of the GEJ or stomach.
2. Patients must be deemed unresectable due to involvement of critical vasculature or adjacent organ invasion. If unresectable, patients must show evidence of disease progression prior to enrollment.
3. Patients with prior surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease unless an interval of > 5 years has elapsed between the primary surgery and the development of metastatic disease. Clinicians should consider biopsy of lesions to establish diagnosis of metastatic disease if there is substantial clinical ambiguity regarding the nature or source of apparent metastases.
4. Prior carboplatin as neoadjuvant or adjuvant therapy will be allowed if >= 6 months from the time of study entry.
5. If patients use aspirin (>325mg/day) or NSAIDS at the time of enrollment, they must have a 10 day washout period prior to beginning protocol treatment.
6. Low molecular weight heparin (or its equivalent, excluding warfarin) will be allowed for treatment of venous thromboembolic events if patients have no evidence of bleeding on full-dose anticoagulation.
7. Patients must have a primary or metastatic lesion measurable in at least one dimension by Modified RECIST criteria (see Section 11.2.3) within 4 weeks prior to entry of study
8. Patients must have ECOG performance status of 0-1
9. Patients must be >= 18 years of age
10. Laboratory values <= 2 weeks prior to randomization:

    * Absolute Neutrophil Count (ANC) >= 1.5 x 109/L (>= 1500/mm3)
    * Platelets (PLT) >= 100 x 109/L (>= 100,000/mm3)
    * Hemoglobin (Hgb) >= 9 g/dL
    * Serum creatinine <= 1.5 x ULN
    * Serum bilirubin <= 1.5 x ULN (<= 3.0 x ULN if liver metastases present)
    * Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) <= 3.0 x ULN (<= 5.0 x ULN if liver metastases present). Note: ERCP or percutaneous stenting may be used to normalize the liver function tests.
11. Life expectancy >= 12 weeks
12. Inclusion and exclusion criteria for DCE-MRI and DWI imaging will be determined by CT scan as part of routine post-chemotherapy imaging. Subjects will be eligible if one liver metastasis is greater than 1 cm in size. Participation in the DCE-MRI and DWI correlate is not required for eligibility.
13. Ability to give written informed consent according to local guidelines

Exclusion Criteria:

1. Disease-Specific Exclusions

   1. Prior chemotherapy for metastatic disease
   2. Prior full field radiotherapy <= 4 weeks or limited field radiotherapy <= 2 weeks prior to enrollment. Patients must have recovered from all therapy-related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease.
   3. Prior biologic or immunotherapy <= 2 weeks prior to registration. Patients must have recovered from all therapy-related toxicities
   4. Prior therapy with anti-VEGF agents
   5. If history of other primary cancer, subject eligible only if she or he has:

      * Curatively resected non-melanomatous skin cancer
      * Curatively treated cervical carcinoma in situ
      * Other primary solid tumor curatively treated with no known active disease present and no treatment administered for the last 3 years
   6. Concurrent use of other investigational agents and patients who have received investigational drugs <= 4 weeks prior to enrollment.
   7. Hypersensitivity to capecitabine, fluorouracil, or any component of the formulation and or a known deficiency of dihydropyrimidine dehydrogenase.
2. General Medical Exclusions

   1. Subjects known to have chronic or active hepatitis B or C infection
   2. History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with study participation or study drug administration or may interfere with the conduct of the study or interpretation of study results
   3. Male subject who is not willing to use adequate contraception upon enrollment into this study and for 6 months following the last dose of second-line treatment
   4. Female subject (of childbearing potential, post-menopausal for less than 6 months, not surgically sterilized, or not abstinent) who is not willing to use an oral, patch or implanted contraceptive, double-barrier birth control, or an IUD during the course of the study and for 6 months following the last dose of second-line treatment
   5. Female subject who is breast-feeding or who has positive serum pregnancy test 72 hours prior to randomization
   6. Pleural effusion or ascites that causes respiratory compromise (>= CTCAE grade 2 dyspnea)
   7. Any of the following concurrent severe and/or uncontrolled medical conditions within 24 weeks of enrollment which could compromise participation in the study:

      * Unstable angina pectoris
      * Symptomatic congestive heart failure
      * Myocardial infarction <= 6 months prior to registration and/or randomization
      * Serious uncontrolled cardiac arrhythmia
      * Uncontrolled diabetes
      * Active or uncontrolled infection
      * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung.
      * Chronic renal disease
      * Acute or chronic liver disease (e.g., hepatitis, cirrhosis)
   8. Patients unwilling to or unable to comply with the protocol
   9. Life expectancy of less than 12 weeks
   10. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
3. Bevacizumab-Specific Exclusions

   1. Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
   2. Any prior history of hypertensive crisis or hypertensive encephalopathy
   3. New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix A)
   4. History of myocardial infarction or unstable angina within 6 months prior to study enrollment
   5. History of stroke or transient ischemic attack within 6 months prior to study enrollment
   6. Known CNS disease, brain metastases.
   7. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
   8. Symptomatic peripheral vascular disease
   9. Evidence of bleeding diathesis or coagulopathy
   10. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
   11. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
   12. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
   13. Serious, non-healing wound, ulcer, or bone fracture
   14. Urine protein >= 2+ on urinalysis dipstick and >= 1.0 gram on 24-hour urine collection
   15. Known hypersensitivity to any component of bevacizumab
   16. History of hemoptysis (bright red blood of ½ teaspoon or more per episode) within 3 months prior to study enrollment.
   17. Current, ongoing treatment with full-dose warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-02; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Kunz, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Indicated participant number is accurate for the number of subjects who started study treatment and completed treatment.
Period: Overall Study
Arm/Group | Bevacizumab+ Carboplatin +Capecitabine
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab+ Carboplatin +Capecitabine
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Tumor progression was assessed according to the Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), presented below.
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Objective Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria.
  Progression-Free Survival is assessed as the number of evaluable participants who were alive without disease progression at 1 year. Participants without out assessment at 12 months will not be included.
Time Frame: 12 months
Population: Those participants who did not receive follow-up at 12 months were considered lost-to-follow-up and not evaluable for progression, and were censored from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab+ Carboplatin +Capecitabine
Number analyzed (Participants) | 28
Participants | 9

2. Secondary Outcome: Adverse Events ≥ Grade 3 and Related to Bevacizumab
Description: Toxicity was assessed as the number of adverse events ≥ Grade 3 and also possibly, probably, or definitely related to bevacizumab. The outcome is reported as the total number of applicable events, and as the number of events that were a hematologic toxicity; a non-hematologic toxicity; which are numbers without dispersion.
Time Frame: 12 months
Population: All participants were included in this analysis.
Measure: Number; unit: Adverse events
Arm/Group | Bevacizumab+ Carboplatin +Capecitabine
Number analyzed (Participants) | 35
Adverse events
  Total Toxicity Events | 18
  Total Hematologic Toxicities | 3
  Total Non-hematologic Toxicities | 15

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) will be assessed from time from the date of enrollment to the date of death due to any cause or the last date the patient was known to be alive (censored observation) at the date of data cutoff for the final analysis. The outcome is presented as the median survival in days with standard deviation.
Time Frame: 7.5 years
Population: Data were available for all participants. Participants remaining alive were censored at last date assessed.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Bevacizumab+ Carboplatin +Capecitabine
Number analyzed (Participants) | 35
Days | 458 (738)

4. Secondary Outcome: Objective (Overall) Therapeutic Response
Description: Tumor response was assessed per the Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions, and assessed by physical measurement; magnetic resonance imaging (MRI); computed tomography (CT), positron emission tomography (PET)-CT; and/or X-rays/radiologic scan. Response was determined based on the criteria below.
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Objective Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria The outcome is provided as the number of participants who achieved each of the defined responses, with objective (overall) response defined as the sum of CR and PR. The outcome is reported as values without dispersion.
Time Frame: 12 months
Population: Data for clinical response was not available for all participants. Response data are only reported for participants for whom response is known.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab+ Carboplatin +Capecitabine
Number analyzed (Participants) | 29
Participants
  Partial Response | 18
  Complete Response (CR) | 0
  Objective Response (OR) = CR + PR | 18
  Stable Disease | 6
  Progressive Disease | 5

5. Secondary Outcome: CEA and CA 19.9 Tumor Response Biomarkers
Description: The detected blood levels for tumor biomarkers CEA and CA 19.9 were to be correlated to the results for progression-fee survival (PFS), with the outcome presented as the median with standard deviation.
Time Frame: 9 weeks
Population: Based on the objective results, it was determined that the any results from tumor biomarker analyses would be of little value, and the measurement for tumor biomarkers in the collected samples were not conducted. Accordingly, there is no data to be analyzed.
Arm/Group | Bevacizumab+ Carboplatin +Capecitabine
Number analyzed (Participants) | 0

6. Secondary Outcome: Vascular Endothelial Growth Factor Tumor Response Biomarker
Description: The detected blood levels for tumor biomarker vascular endothelial growth factor (VEGF) were to be correlated to the results for progression-fee survival (PFS), with the outcome presented as the median with standard deviation.
Time Frame: 9 weeks
Population: Studies published during the conduct of this study demonstrated that this assessment was not useful, and the samples were not collected. Accordingly, there is no data to be analyzed.
Arm/Group | Bevacizumab+ Carboplatin +Capecitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 7.5 years
Arm/Group | Bevacizumab+ Carboplatin +Capecitabine
All-Cause Mortality (participants affected / at risk) | 31/35
Serious Adverse Events (participants affected / at risk) | 35/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab+ Carboplatin +Capecitabine (N=35)
Nausea (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Obstruction gastric (Gastrointestinal disorders) | 3 (3)
Death NOS (General disorders) | 4 (4)
Multi-organ failure (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Other, pulmonary embolism (Vascular disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Plural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Other, disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27 (27)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab+ Carboplatin +Capecitabine (N=35)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 26 (42)
Leukocytosis (Blood and lymphatic system disorders) | 23 (32)
Neutrophil count decreased (Blood and lymphatic system disorders) | 23 (36)
Platelet count decreased (Blood and lymphatic system disorders) | 30 (45)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 11 (14)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 7 (9)
Hypotension (Vascular disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Fatigue (General disorders) | 29 (46)
Chills (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Weight loss (Investigations) | 5 (5)
Sweating (hyperhidrosis, diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 15 (22)
Rash (Infections and infestations) | 17 (29)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Infections and infestations -Other, specify desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 15 (17)
Nausea (Gastrointestinal disorders) | 25 (31)
Vomiting (Gastrointestinal disorders) | 15 (16)
Diarrhea (Gastrointestinal disorders) | 18 (22)
Dehydration (Metabolism and nutrition disorders) | 6 (7)
Mucositis (Gastrointestinal disorders) | 11 (11)
Constipation (Gastrointestinal disorders) | 11 (11)
Gastrointestinal disorders -Other, specify Enteritis (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 6 (6)
Bloating (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (19)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 7 (7)
Renal and urinary disorders - Other, specify Hemorrhage Urinary (Renal and urinary disorders) | 6 (6)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 2 (2)
Periodontal disease (Infections and infestations) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (7)
Proteinuria (Renal and urinary disorders) | 10 (15)
Aspartate aminotransferase increased (Investigations) | 15 (16)
hypoalbuminemia (Metabolism and nutrition disorders) | 10 (13)
Alkaline phosphatase (Investigations) | 10 (12)
Alanine aminotransferase increased (Investigations) | 9 (10)
Creatinine increased (Investigations) | 6 (6)
Hyponatremia) (Metabolism and nutrition disorders) | 5 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Lipase increased (Investigations) | 1 (1)
Joint range of motion decreased, upper extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 4 (4)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 9 (9)
Ataxia (Nervous system disorders) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1)
Watering eyes (Eye disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Pain- Joint (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Renal and urinary disorders -Other, specify Urethera pain (Renal and urinary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (8)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory, thoracic andmediastinal disorders - Other, specify paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Libido (Psychiatric disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT00780494/Prot_SAP_000.pdf